CLINICAL TRIAL: NCT04022954
Title: HD Mapping Observational Study - Asia Pacific
Brief Title: HD Mapping of Atrial Fibrillation in Asia Pacific
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: CRD975
Record Dates: First submitted 2019-06-29; First posted 2019-07-17 (Actual); Results first posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2023-10

CONDITIONS: Paroxysmal Atrial Fibrillation; Persistent Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Inquiry™ AFocusII™ Double Loop: The Inquiry™ AFocus™ catheters are for recording intracardiac signals and cardiac stimulation during diagnostic electrophysiological studies. The Inquiry™ AFocus™ catheters are for use in mapping atrial regions of the heart.
  Interventions: Device: Catheter ablation
- Advisor™ HD Grid, Sensor Enabled™: The Advisor™ HD Grid Mapping Catheter, Sensor Enabled™, is indicated for multiple electrode electrophysiological mapping of cardiac structures in the heart with recording or stimulation only. This catheter is intended to obtain electrograms in the atrial and ventricular regions of the heart.
  Interventions: Device: Catheter ablation

INTERVENTIONS:
Device: Catheter ablation — Inquiry AFocusII Double Loop and Advisor HD Grid, Sensor Enabled

SUMMARY:
The aim of this study is to quantify and characterize the outcomes of radiofrequency (RF) ablation after, and the utility of, electroanatomical mapping with the market-released HD mapping catheters Inquiry™ AFocusII™ Double Loop and Advisor™ HD Grid, Sensor Enabled™ with the EnSite Cardiac Mapping System and the EnSite Automap module in subjects with AF in the real-world environment of the Asian population.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must provide written informed consent for study participation and willing and able to comply with the protocol described evaluations and follow up schedule
2. Subject must be over 18 years of age. (In Japan, the subject must be of 20 years of age or older)
3. Subject is diagnosed with AF as defined by:

   * Documented symptomatic paroxysmal AF defined as AF that terminates spontaneously or with intervention within 7 days of onset
   * Documented symptomatic persistent AF defined as continuous atrial fibrillation that is sustained beyond 7 days but less than 12 months
4. Subject is indicated for cardiac electroanatomical mapping and RF ablation procedure to treat AF
5. Subject is planned to have electroanatomical mapping performed with the HD mapping catheters under investigation

Exclusion Criteria:

1. Previous ablation or surgery in the left atria
2. Implanted left atrial appendage occluder
3. Implanted mitral or tricuspid valve replacement
4. Implanted cardiac defibrillator (ICD)
5. Participation in another clinical investigation that may confound the results of this study
6. Pregnant or nursing
7. Presence of other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements, or impact the scientific soundness of the clinical investigation results.
8. Life expectancy less than 12 months

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The analysis population used for all endpoints will include all subjects who have signed the Informed Consent Form and have undergone the electroanatomical mapping procedure using one of the specified HD mapping catheters and received RF ablation as specified in the protocol. If any device used during the procedure is used off-label, the subject will be excluded from non-safety related endpoint analysis and any additional evaluations
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-09-11 (Actual); Primary Completion 2021-08-13 (Actual); Study Completion 2021-08-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Ruffner, PhD, Study Director — EP Program Director
Locations (15):
- China (2):
  - Sir Run Run Shaw Hospital, Hangzhou
  - The Second Affiliated Hospital of Xian Jiaotong University, Xi'an
- Prince of Wales Hospital, Hong Kong, Hong Kong
- Japan (8):
  - Kokura Memorial Hospital, Kitakyushu-shi, Fukuoka
  - University of Tsukuba Hospital, Tsukuba, Ibaraki
  - Yokosuka Kyosai Hospital, Kanagawa
  - Kyoto University Hospital, Kyoto
  - Ogaki Municipal Hospital, Ōgaki
  - Saga University Hospital, Saga
  - Kitasato University Hospital, Sagamihara
  - Kyorin University Hospital, Tama
- South Korea (2):
  - Korea University Anam Hospital, Seoul
  - Severance Hospital, Seoul
- Taiwan (2):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Taipei Veterans General Hospital (VGH), Taipei

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 201 consented patients, 200 met the protocol definition for subject enrollment (including written informed consent AND HD mapping catheter inserted) and were considered enrolled in the study. One consented subject was a screen failure due to operator choice of a different system (non-study device) prior to procedure. Because a study-specified HD mapping catheter was not inserted, this patient was withdrawn prior to the Baseline Visit as a consented non-enrolled screen failure.
Groups:
- Electroanatomical Mapping With HD Mapping Catheter: Subjects underwent electroanatomical mapping procedure using one of the specified HD mapping catheters and received RF ablation as specified in the protocol.
Period: Consented to Completed Procedure
Arm/Group | Electroanatomical Mapping With HD Mapping Catheter
Started | 201
Completed | 200
Not Completed | 1
Not completed — Consented Screen Failure | 1
Period: Completed 12-month Follow-up
Arm/Group | Electroanatomical Mapping With HD Mapping Catheter
Started | 200
Completed | 192
Not Completed | 8
Not completed — Lost to Follow-up | 5
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Electroanatomical Mapping With HD Mapping Catheter
Number analyzed (Participants) | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.0 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62
  Male | 138
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 200
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  South Korea | 37
  Hong Kong | 11
  China | 6
  Japan | 101
  Taiwan | 45
Height [Mean (Standard Deviation); unit: centimeters] — Population: No baseline height from one subject.
  centimeters
    number analyzed (Participants) | 199
    (all) | 166.0 (9.8)
Weight [Mean (Standard Deviation); unit: kilograms] — Population: No baseline weight from one subject.
  kilograms
    number analyzed (Participants) | 199
    (all) | 69.0 (14.6)
Heart Rate on ECG [Mean (Standard Deviation); unit: bpm] — Population: No Heart rate on ECG data at baseline for 5 subjects.
  bpm
    number analyzed (Participants) | 195
    (all) | 72.9 (20.3)
Rhythm on ECG [Count of Participants; unit: Participants] — Population: Rhythm on ECG is only available for 196/200 enrolled subjects.
  Participants
    Sinus Rhythm: number analyzed (Participants) | 196
    Sinus Rhythm | 127
    Atrial Fibrillation: number analyzed (Participants) | 196
    Atrial Fibrillation | 37
    Typical Atrial Flutter (CTI dependent): number analyzed (Participants) | 196
    Typical Atrial Flutter (CTI dependent) | 4
    Atypical Atrial Flutter (non-CTI dependent): number analyzed (Participants) | 196
    Atypical Atrial Flutter (non-CTI dependent) | 7
    Sinus rhythm with PVC: number analyzed (Participants) | 196
    Sinus rhythm with PVC | 2
    A-paced with intrinsic conduction: number analyzed (Participants) | 196
    A-paced with intrinsic conduction | 1
    Sinus rhythm with PAC: number analyzed (Participants) | 196
    Sinus rhythm with PAC | 1
    Sinus bradycardia: number analyzed (Participants) | 196
    Sinus bradycardia | 14
    Other: number analyzed (Participants) | 196
    Other | 3
History of Heart Failure [Count of Participants; unit: Participants] — Population: Analysis population for New York Heart Association (NYHA) heart failure classes only includes those subjects with a history of heart failure. NYHA class is a standardized, widely accepted measure of heart failure symptom severity (see for example CW Yancy et al., Circulation, 128 (2013), pp. e240-e327). A patient can be evaluated by a cardiologist (heart doctor) to determine if heart failure symptoms are present and to classify the severity from Class I (least severe) to Class IV (most severe).
  Participants
    History of Heart Failure | 15
    Class I: number analyzed (Participants) | 15
    Class I | 6
    Class II: number analyzed (Participants) | 15
    Class II | 3
    Class III: number analyzed (Participants) | 15
    Class III | 1
    Class IV: number analyzed (Participants) | 15
    Class IV | 0
    Not Evaluated: number analyzed (Participants) | 15
    Not Evaluated | 5
Cardiomyopathy [Count of Participants; unit: Participants] | 6
Valvular Heart Disease [Count of Participants; unit: Participants] | 17
Hypertension [Count of Participants; unit: Participants] | 105
Stroke/TIA/Thromboembolism [Count of Participants; unit: Participants] — Population: No history of stroke/TIA/thromboembolism collected at baseline for 4 subjects.
  Participants
    number analyzed (Participants) | 196
    (all) | 15
Conduction Disease [Count of Participants; unit: Participants] | 8
Arrhythmia History [Count of Participants; unit: Participants]
  Paroxysmal | 169
  Persistent | 23
  Longstanding Persistent | 6
  Typical Flutter | 21
  Atypical Flutter | 3
  Type Unknown Flutter | 5
  Atrial Tachycardia | 2
  Multifocal AT | 0
  AVRT/Accessory Pathway | 0
  AVNRT | 1
  Ischemic Ventricular Tachycardia | 0
  Non-ischemic ventricular tachycardia | 0
  Idiopathic Ventricular Tachycardia | 1
  PVCs | 8
Indication for this procedure [Count of Participants; unit: Participants]
  Symptomatic Paroxysmal AF | 165
  Symptomatic Persistent AF | 35
History of Class I or III AAD use [Count of Participants; unit: Participants] | 155

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Acute Success of RF Ablation After Electroanatomical Mapping With HD Mapping Catheters.
Description: The rate of acute success was defined as the proportion of subjects who receive HD mapping and RF energy delivery resulting in acute termination of clinical arrhythmia, defined by termination to SR (or AT if being treated for PersAF) or non-inducibility of clinical arrhythmia after ablation (cardioversion allowed prior to inducibility attempt). This measure is presented here as the number of participants with acute success, and the associated percentage of subjects (proportion * 100%) with acute success is also displayed as the result of an automatic calculation.
Time Frame: End of Procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Electroanatomical Mapping With HD Mapping Catheter
Number analyzed (Participants) | 200
Participants | 173

2. Primary Outcome: Number of Participants With Clinical Long-Term Success
Description: Freedom from all atrial arrhythmias (AF/AFL/AT) greater than 30 seconds (as documented by 24-hr Holter at 12-month follow-up) and on or off class I/III AADs. This measure is presented here as the number of participants, and the associated percentage of subjects (proportion * 100%) is also displayed as the result of an automatic calculation.
Time Frame: 12 months post-procedure
Population: Overall Number of Participants Analyzed is the number of subjects that have completed a 24-hour Holter at 12 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Electroanatomical Mapping With HD Mapping Catheter
Number analyzed (Participants) | 182
Participants | 168

3. Primary Outcome: Number of Participants With AAD-Free Long-Term Success
Description: Freedom from all atrial arrhythmias (AF/AFL/AT) greater than 30 seconds (as documented by 24-hr Holter at 12-month follow-up) and off all class I/III AADs. This measure is presented here as the number of participants, and the associated percentage of subjects (proportion * 100%) is also displayed as the result of an automatic calculation.
Time Frame: 12-month post-procedure
Population: Overall Number of Participants Analyzed is the number of subjects that have completed a 24-hour Holter at 12 months or have documented Class I or III AAD use between the end of the blanking period and 12-months.
Measure: Count of Participants; unit: Participants
Arm/Group | Electroanatomical Mapping With HD Mapping Catheter
Number analyzed (Participants) | 189
Participants | 104

4. Secondary Outcome: Overall Procedure Time
Description: Defined as time from initial catheter insertion to final catheter removal. This is one measure of the amount of time it took for the physician to use invasive tools (catheters) during the procedure to investigate, diagnose, and treat the participant's heart condition.
Time Frame: During Procedure
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Electroanatomical Mapping With HD Mapping Catheter
Number analyzed (Participants) | 200
minutes | 152.9 (50.3)

5. Secondary Outcome: Radiofrequency (RF) Time
Description: Defined as duration of time radiofrequency energy is delivered. This is a measure the amount of time the physician was actively applying treatment to the heart to treat the participant's heart condition.
Time Frame: During Procedure
Population: Overall Number of Participants Analyzed is the number of subjects with available data for this outcome.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Electroanatomical Mapping With HD Mapping Catheter
Number analyzed (Participants) | 199
minutes | 35.9 (14.3)

6. Secondary Outcome: Fluoroscopy Time
Description: Defined as total time subject is exposed to fluoroscopy. Fluoroscopy is a type of medical imaging that uses x-rays. This imaging is used by the physician to facilitate a safe and effective procedure. Less fluoroscopy time may help reduce the risk of issues related to x-ray exposure, however other factors such as fluroscopy intensity (not measured in this study) may also be important.
Time Frame: During Procedure
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Electroanatomical Mapping With HD Mapping Catheter
Number analyzed (Participants) | 200
minutes | 38.7 (31.2)

7. Secondary Outcome: Mapping Time Associated With Mapping Arrhythmia
Description: Defined as the total cumulative mapping time and mapping time for the creation of each map (including any new or retrospective map created with Manual, AutoMap, and TurboMap mapping). As part of an ablation procedure to treat atrial fibrillation, some physicians create a map of the heart's electrical activity. The information in the map may be used by the physician to plan the treatment strategy. Mapping time provides a measure of how much time the physician spent creating, updating, and analyzing maps during the procedure. A short mapping time is not necessarily better or worse than a long mapping time, as other factors such as the amount and type of information gathered may also affect how useful the map is to the physician.
Time Frame: During Procedure
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Electroanatomical Mapping With HD Mapping Catheter
Number analyzed (Participants) | 200
minutes | 76.3 (63.0)

8. Secondary Outcome: Number of Mapping Points Collected
Description: Defined as total number of mapping points collected for the creation of each map. As part of an ablation procedure to treat atrial fibrillation, some physicians create a map of the heart's electrical activity. The information in the map may be used by the physician to plan the treatment strategy. Number of mapping points collected is a measure of how much information was collected. A small number of mapping points collected is not necessarily better or worse than a large number of points, as other factors such as the amount of time spent and type of information gathered may also affect how useful the map is to the physician.
Time Frame: During Procedure
Measure: Mean (Standard Deviation); unit: mapping points
Units Other Than Participants: Number of Maps
Arm/Group | Electroanatomical Mapping With HD Mapping Catheter
Number analyzed (Participants) | 200
Number analyzed (Number of Maps) | 424
mapping points | 9828.8 (7192.1)

9. Secondary Outcome: Number of Mapping Points Used
Description: Defined as the total number of mapping points used in each map. As part of an ablation procedure to treat atrial fibrillation, some physicians create a map of the heart's electrical activity. The information in the map may be used by the physician to plan the treatment strategy. Number of mapping points collected is a measure of how much information was collected, while number of mapping points used is a measure of how many such points were considered useful. A small number of mapping points used is not necessarily better or worse than a large number of points, as other factors such as the amount of time spent and type of information gathered may also affect how useful the map is to the physician.
Time Frame: During Procedure
Measure: Mean (Standard Deviation); unit: Mapping Points
Units Other Than Participants: Mapping Points
Arm/Group | Electroanatomical Mapping With HD Mapping Catheter
Number analyzed (Participants) | 200
Number analyzed (Mapping Points) | 424
Mapping Points | 1962.4 (1100.0)

10. Secondary Outcome: Number of Used Mapping Points Per Minute
Description: Defined as the total number of mapping points used divided by the relative mapping time. As part of an ablation procedure to treat atrial fibrillation, some physicians create a map of the heart's electrical activity. The information in the map may be used by the physician to plan the treatment strategy. Mapping time is a measure of how much time the physician spent collecting, updating, and analyzing the information in the map. Number of mapping points collected is a measure of how much information was collected, while number of mapping points used is a measure of how many such points were considered useful. The number of used mapping points per minute is a measure of how efficient the mapping process is. A larger number of used mapping points per minute may be associated with a more efficient mapping process. Mapping efficiency may be of interest to a physician, however other factors such as the type of information gathered may also be of interest.
Time Frame: During Procedure
Measure: Mean (Standard Deviation); unit: Number of Mapping Points/Minute
Units Other Than Participants: Number of Maps
Arm/Group | Electroanatomical Mapping With HD Mapping Catheter
Number analyzed (Participants) | 200
Number analyzed (Number of Maps) | 424
Number of Mapping Points/Minute | 231.7 (126.9)

11. Secondary Outcome: Substrate Characteristics Identified
Description: For each type of arrhythmogenic substrate this will be defined as the frequency of substrate type identified in cases that attempted to identify the specific substrate. As part of an ablation procedure to treat atrial fibrillation, some physicians create a map of the heart's electrical activity or use other tests to characterize the state, function, or health of certain areas of the heart tissue, and to localize certain areas that may be problematic (substrate). These localized characteristics may provide information to the physician that could be used to treat the participant's heart condition. This outcome measure lists common substrate characteristics and the number of subjects for which the characteristic was found or otherwise used as part of the treatment plan.
Time Frame: During Procedure
Population: The analysis population is the number of subjects in which the substrate type was searched for
Measure: Count of Participants; unit: Participants
Arm/Group | Electroanatomical Mapping With HD Mapping Catheter
Number analyzed (Participants) | 200
Participants
  Low Voltage | 181
  Fibrosis/Scar: number analyzed (Participants) | 57
  Fibrosis/Scar | 40
  Focal Impulses: number analyzed (Participants) | 2
  Focal Impulses | 1
  Rotors: number analyzed (Participants) | 0
  Rotors | 0
  CFE: number analyzed (Participants) | 4
  CFE | 4
  Other: number analyzed (Participants) | 4
  Other | 4
  Both Low Voltage and Fibrosis/Scar: number analyzed (Participants) | 57
  Both Low Voltage and Fibrosis/Scar | 40

12. Secondary Outcome: Ablation Strategy(s) Used
Description: Defined by both the type of map used to define ablation strategy and the frequency each ablation strategy/target was used by physicians. A physician may use one or more strategies to treat the participant's heart condition, including selectively burning (ablating) certain areas of the heart. This outcome measure lists common ablation strategies and the number of participants that received treatment based on each strategy.
Time Frame: During Procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Electroanatomical Mapping With HD Mapping Catheter
Number analyzed (Participants) | 200
Participants
  Any PVI | 200
  PVI (Common Left) | 110
  PVI (Common Right) | 100
  PVI (LSPV) | 93
  PVI (LIPV) | 92
  PVI (RSPV) | 98
  PVI (RIPV) | 99
  Any Non-PVI | 148
  Eustachian Ridge | 1
  Mitral Isthmus | 1
  LAA Isolation | 2
  Fossa Ovalis | 1
  Roof | 22
  Christa Terminalis | 2
  LAA Focal Ablation | 6
  Coronary Sinus | 1
  CTI | 127
  Posterior Wall Isolation | 10
  SVC Isolation | 26
  Ligament of Marshall | 23
  Box isolation of fibrotic areas | 4
  CFE | 1
  Other | 6

13. Other Pre Specified Outcome: Number of Participants With Adverse Events
Description: Adverse events include any device-, procedure-, or death-related events
Time Frame: through study completion, an average of 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Electroanatomical Mapping With HD Mapping Catheter
Number analyzed (Participants) | 200
Participants | 10

14. Other Pre Specified Outcome: Number of Subjects With Repeat Ablations
Description: Rate of repeat ablations was defined as proportion of subjects with an additional ablation procedure to treat indicated cardiac arrhythmia (outside blanking period, if applicable). This measure is presented here as the number of participants, and the associated percentage of subjects (proportion * 100%) is also displayed as the result of an automatic calculation.
Time Frame: 12-months post-procedure
Population: Overall Number of Participants Analyzed is the number of subjects that have either completed 12 months of follow up, or not completed 12 months of follow up but have experienced an additional ablation procedure to treat indicated cardiac arrhythmia outside of the blanking period.
Measure: Count of Participants; unit: Participants
Arm/Group | Electroanatomical Mapping With HD Mapping Catheter
Number analyzed (Participants) | 192
Participants | 7

15. Other Pre Specified Outcome: Change in Quality of Life (QoL): EQ-5D-5L VAS Score
Description: Defined as change in quality of life score assessed by the validated QoL survey, EQ-5D-5L. The EQ-5D-5L is a descriptive system comprised of five questions related to mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each question has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  EQ-5D-5L EQ VAS scores range from 0 (worst) to 100 (best). A positive change indicates an improvement.
Time Frame: 12-months post-procedure
Population: The overall number of participants considered for analysis for the quality of life metrics was the 200 enrolled subjects. The number analyzed for each individual metric includes the subjects with data at both baseline and the timepoint of interest (6-months or 12-months). Of 200 enrolled subjects, 197 had available data both at baseline and 6 months. Of 200 enrolled subjects, 192 subjects had available data both at baseline and 12 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Electroanatomical Mapping With HD Mapping Catheter
Number analyzed (Participants) | 200
score on a scale
  VAS Score Change from Baseline to 6-months: number analyzed (Participants) | 197
  VAS Score Change from Baseline to 6-months | 6.7 (14.3)
  VAS Score Change from Baseline to 12-months: number analyzed (Participants) | 192
  VAS Score Change from Baseline to 12-months | 5.4 (17.1)

ADVERSE EVENTS:
Time Frame: 12 months
Description: Adverse events collected were only those considered related to either the ablation catheter or the ablation procedure by the investigator or resulted in death.
  All-Cause Mortality: all anticipated and unanticipated deaths due to any cause. Serious Adverse Events: all anticipated and unanticipated serious adverse events related (or possibly related) to procedure or device.
  Other Adverse Events: anticipated and unanticipated non-serious events related to procedure or device.
Arm/Group | Electroanatomical Mapping With HD Mapping Catheter
All-Cause Mortality (participants affected / at risk) | 0/200
Serious Adverse Events (participants affected / at risk) | 5/200
Other Adverse Events (participants affected / at risk) | 5/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Electroanatomical Mapping With HD Mapping Catheter (N=200)
Cerebrovascular Accident/Stroke (Nervous system disorders) | 2
Pericardial Effusion (Cardiac disorders) | 2
Retroperitoneal Hematoma (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Electroanatomical Mapping With HD Mapping Catheter (N=200)
Bleeding/Anemia (Vascular disorders) | 1
Fever (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia (Infections and infestations) | 1
Vascular Access Complications (Vascular disorders) | 1
Vascular Bleeding/Local Hematomas/Ecchymosis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
First publication of study results will be made as a joint multi-center publication with investigators from all sites contributing data. Institutions may publish data and results individually from its site after any of the following (1) a multi-center publication is published, (2) no multicenter publication is submitted within eighteen months after closures of the Study at all sites or (3) sponsor confirms in writing there will be no multi-center publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-06): https://cdn.clinicaltrials.gov/large-docs/54/NCT04022954/Prot_SAP_000.pdf